CLINICAL TRIAL: NCT05726006
Title: Invasive Group B Streptococcus Disease Burden and Its Antimicrobial Resistance in Malaysia Among Non-pregnant Adults: a Prospective Observational Protocol Study
Brief Title: Invasive Group B Streptococcus Disease Burden and Its Antimicrobial Resistance in Malaysia Among Non-pregnant Adults.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, AbdulRahman Mansoor Mohammed Muthanna, Research Assistant, Universiti Putra Malaysia
Other Study IDs: UPM-PhD AbdulRahman
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Invasive Infection; Diabetic Foot; Immunocompromised Patients; Group B Streptococcal Infections
MeSH Terms: conditions — Diabetic Foot; Streptococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bacteria strains will be isolated, cultivated, and identified in the hospital laboratories. Sterile samples will be cultured using automated blood culture systems.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-pregnant adult patients with group B streptococcal infection: all non-pregnant adult patients from the selected hospitals whom group B streptococcus will be isolated from their clinical samples from sterile sites.
  Interventions: Other: No Intervention in This study

INTERVENTIONS:
Other: No Intervention in This study — No Intervention in This study

SUMMARY:
Group B Streptococcus (GBS) infection is a potential aetiology of meningitis and septicemia in neonates, pregnant women and non-pregnant adults. Because the GBS disease burden is unknown in Malaysia, it is unlikely to receive much attention. This study aims to determine the prevalence of group B streptococcus isolated from non-pregnant adults, the Incidence, case-fatality ratio, antimicrobial susceptibility patterns, serotyping, genotyping and detection of the GBS virulence and pili genes from six major hospitals in Peninsular Malaysia.

DETAILED DESCRIPTION:
This multicentre, prospective, observational study will be conducted in six major tertiary hospitals in Malaysia among Non-Pregnant Adults. At the same time, a retrospective study will be conducted on the selected hospitals to determine GBS strains and data. GBS isolates will be subjected to phenotyping, serotyping using Multiplex PCR, antimicrobial susceptibility testing and detection of GBS virulence and pilus genes. Seven housekeeping genes will be sequenced internally to perform multi-locus sequence typing (MLST). Findings from the study will contribute to improving clinical practice to diagnose and prevent GBS disease on time. The prudent use of antibiotics will be encouraged by monitoring antimicrobial resistance.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adult patients
* patients with group B streptococcus infection
* The clinical samples isolated from sterile sites (blood, cerebrospinal fluid, internal tissue, pus aspirate, peritoneal dialysis fluid, bone biopsy, skin biopsy and bone marrow).

Exclusion Criteria:

* Repeated group B streptococcus that is isolated from the same patients in the same admission
* Non-sterile site isolates (Urine, Vaginal swab)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consist of all non-pregnant adult patients from the selected hospitals whom group B streptococcus were isolated from their clinical samples from sterile sites (blood, cerebrospinal fluid, internal tissue, pus aspirate, peritoneal dialysis fluid, bone biopsy, skin biopsy and bone marrow). Repeated GBS that is isolated from the same patients in the same admission and non-sterile site isolates will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
To examine the prevalence of invasive GBS illness among non-pregnant people in Malaysia. | 18 months
  . The researcher will verify the participants' medical records. Data on demographic data, clinical information, and information about the treatment and diagnosis initiated by the attending physician will be collected from patient's medical records from the selected hospitals.
To examine the prevalence of antibiotic resistance of invasive GBS isolates among non-pregnant people in Malaysia. | 2 months
  The disc diffusion (Kirby-Bauer) method will be used to determine the antimicrobial susceptibility of the GBS isolates to penicillin, ampicillin, clindamycin, erythromycin, vancomycin, tetracycline, azithromycin, ceftriaxone, cefotaxime, cefepime, ofloxacin, chloramphenicol, linezolid (Oxoid, Basingstoke, UK). Meanwhile, the E-test method will be used to determine the minimal inhibitory concentrations (MIC) of resistant strains. The diameter of inhibition zones will be measured, and MIC will be read based on the recently stated CLSI guideline (Clinical and Laboratory Standards Institute (CLSI), 2022).

SECONDARY OUTCOMES:
Detection of GBS Virulence and Pilus Genes | 3 months
  GBS virulence (cfb, cylE, lmb, scpB, hylB, rib, fbsA, fbsB, spb1, bca and bac) and pili genes (PI-1, PI-2a and PI-2b) will be amplified using PCR that performed on a BioRadMyCyclerTM Thermal Cycler (BioRad, Massachusetts, USA) using the primers and running conditions published previously
Detection of Capsular polysaccharides types of GBS using Multiplex PCR | 3 months
  GBS capsular serotypes will be deduced by the multiplex PCR method. Ten serotypes (Ia, Ib and II - IX) will be determined by targeting the cps gene cluster, including cpsL, cpsG, cpsJ-Ib, cpsJ-2, cpsG-3-6, cpsJ-4, cpsN-5, cpsI-6, cpsI-7, cpsJ-8, and cpsI-9 genes using published primers according to the study by Imperi et al. (2010).
Detection of Sequence Type (ST) | 3 mnths
  Multi-locus sequence typing (MLST) will be performed by sequencing the internal fragments of seven housekeeping genes (ashP, pheS, atr, glnA, sdhA, glcK and tkt), as previously described (Jones et al., 2003). The sequences of the seven housekeeping genes will be trimmed and aligned using Molecular Evolutionary Genetics Analysis version 7 (MEGA 7) software according to known alleles base pair as described in the MLST database website (http://pubmlst.org/) in order to determine the allelic number and sequence type (ST).

CONTACTS AND LOCATIONS:
Overall Officials: AbdulRahman Muthanna, PhD, Principal Investigator — FACULTY OF MEDICINE AND HEALTH SCIENCES, UNIVERSITI PUTRA MALAYSIA (UPM)
Locations (1):
- Faculty of Medicine and Health Sciences, Serdang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol